CLINICAL TRIAL: NCT00282451
Title: Comparison of Biphasic Insulin Aspart 30 Twice Daily With Biphasic Insulin Aspart 30 Twice Daily Plus Lunchtime Injection of Insulin Aspart, in Combination With or Without Metformin (for Both Treatment Groups) in Subjects With Type 2 Diabetes. A Multi-center, Randomized, Open-labeled, Two-armed Parallel Group Trial in Subjects With Type 2 Diabetes Previously Treated With Conventional Biphasic Human Insulin 30/70
Brief Title: Effect of Biphasic Insulin Compared to Biphasic Insulin Combined With Insulin Aspart, With or Without Metformin in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3024
Record Dates: First submitted 2006-01-25; First posted 2006-01-26 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Drug: insulin aspart

SUMMARY:
This trial is conducted in Africa and Middle East. The objective of the study is to compare glycemic control of Biphasic insulin Aspart 30 twice daily with Biphasic insulin Aspart 30 twice daily plus Insulin Aspart, both insulin treatments with or without metformin, in subjects with type 2 diabetes, previously treated with Biphasic Human Insulin 30/70.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic subjects
* Current treatment with Biphasic Human Insulin 30/70 twice daily alone or in combination with any oral hypoglycaemic agent for at least 3 months prior to entering the trial
* HbA1c at least 12%
* Willing and able to perform self blood glucose monitoring (SMBG)

Exclusion Criteria:

* History of drug or alcohol dependence
* Receipt of any investigational drug within the last month prior to this trial
* Anticipated change in dose of prescription medication, which may influence glucose regulation (Mono Amino Oxidase-inhibitors, non selective beta-adrenergic agents, anabolic steroids and systemic glucocorticoids)
* Severe uncontrolled hypertension
* Recurrent severe hypoglycemia as judged by investigator
* Any disease or condition, which the Investigator feels, would interfere with the trial

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2006-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | At Visit 6 (14 weeks)

SECONDARY OUTCOMES:
Postprandial glucose concentration increments (calculated based on 7-point blood glucose profiles)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- Egypt (2):
  - Novo Nordisk Investigational Site, Aghakhan
  - Novo Nordisk Investigational Site, Giza
- Saudi Arabia (2):
  - Novo Nordisk Investigational Site, Jeddah
  - Novo Nordisk Investigational Site, Riyadh

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com